CLINICAL TRIAL: NCT04982523
Title: Development and Evaluation of an Online Mental Health Program for Traumatized Female College Students: A Randomized Controlled Trial
Brief Title: Online Mental Health Program for Female College Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CHA University (Other)
Responsible Party: Principal Investigator, Lee, Kyunghyun, Assistant professor, CHA University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Nursing001
Record Dates: First submitted 2021-07-21; First posted 2021-07-29 (Actual); Last update posted 2021-07-29 (Actual); Status verified 2021-07

CONDITIONS: Post Traumatic Stress Disorder
Keywords: Stress Disorders, Post-Traumatic; Depression; Internet-Based Intervention; Cognitive Behavioral Therapy
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Online Mental Health Program Group (Experimental): The online mental health program of 8 sessions is provided. Data collection was collected pre-, post-, and one month after the program.
  Interventions: Behavioral: Online Mental Health Program
- Control Group (No Intervention): Data collection was collected three times for three months. No intervention was provided during the study.
  If they wanted, they were provided the online mental health program same as the experimental group after data collection.

INTERVENTIONS:
Behavioral: Online Mental Health Program — The proposed program consisted of eight sessions conducted twice per week, consisting of 5 minutes of introductory material, 12-15 minutes of main content, and 5 minutes of concluding content. The main content intended to improve the control processes and each of the four adaptive modes of the RAM. The eight sessions were uploaded on the web. Links and passwords for each session were provided to the participants through SNS. The program was accessible from any electronic device with Internet access
  Arms: Online Mental Health Program Group

SUMMARY:
Late adolescence and early adulthood are the most exposed to trauma. College students exposed to trauma may experience depression, anxiety, stress, and difficulties adapting to college life.

Depression symptoms are the most common reactions that people experience after traumatic experiences. Depression also harms college students reactions that people experience after traumatic experiences. It is difficult for people who are depressed to meet their social function.

Trauma also has adverse physical effects, including dysfunction of the hypothalamus and adrenal axis, lowering blood cortisol levels. As a result, the body's immune system is disturbed, leaving people more exposed to diseases and experiencing more pain and fatigue.

In particular, women are more vulnerable to PTSD than men. Women with post-traumatic stress and depression are also more likely to be exposed to several diseases. Moreover, when traumatized female college students experience life stress, it worsens their mental health and interferes with their studies.

Cognitive behavioral therapy is the most effective content composition method for trauma intervention. CBT should be improved by helping to reduce PTSS and depression and managing various aspects of life, such as nutrition, activity, and rest.

One major advantage of online programs is that they do not face any time or space constraints, and they are also less expensive than face-to-face programs. More importantly, online programs can reduce psychological barriers to participation. This is especially important for women who are more likely to feel shame and stigma about interpersonal traumas, such as those arising from relationships and sexual trauma, which are obstacles to their access to face-to-face programs. College students can easily access online programs because of their familiarity with the Internet, so the programs can be immediately available in response to crises without requiring them to expose personal information to unfamiliar therapists.

In this study, the interventions program was based on the Roy Adaptation Model to address post-traumatic physical and mental health problems among female college students in Korea.

Hypothesis

* The post-traumatic stress scores, depressive symptom scores of participants who access the program will decrease more than those who do not.
* The functional health scores, college adaptation scores of participants who access the program will increase more than those who do not.

DETAILED DESCRIPTION:
1. Study Design This study used a randomized control group pretest-posttest design to verify the effectiveness of the proposed program.
2. Participants & Recruitment Initial participants were recruited from eight universities in Korea through advertisements on SNS and bulletin boards at the university. Applicants indicated their interest in the study by contacting the research director via SNS, email, or SMS. The research director sent a reply message with the research information and an initial screening survey link. The applicants were initially screened for post-traumatic stress and depression. For inclusion, the participants had to be female college students between 19 and 29 years with a traumatic experience and post-traumatic stress symptom scores of 22-66, which is a cutoff that can be diagnosed as post-traumatic stress disorder; anything above 66 is a severe post-traumatic stress disorder condition that cannot be suitably addressed in this study (Eun, 2005; Lee et al., 2018).

   The following participants were excluded: those who experienced childhood sexual abuse; those who had experienced violent conflict or war, including North Korean defectors; and those who had a post-traumatic stress score greater than 66 points. According to a prior study, those who experienced childhood sexual abuse, war, or civil war are at a higher risk of suicide attempts. Therefore, they were excluded because their profiles did not match the purpose of this study (Hirai & Clum, 2005).

   The number of subjects for this study was calculated by G × power using a calculating power of 0.8 for the replicate measurement variance analysis, a medium effect size of 0.25, and a significance level of .05 (Cohen, 1988), resulting in a total of 28 people. Fifty-eight people will be recruited, taking into account the dropout rate of 30%.
3. Procedure The experimental group's pre- and post-outcome measures were collected at pre-treatment, post-treatment, and 1-month follow-up. Data were collected from the control group three times for three months. After the three surveys, the control group was provided the same program as the experimental group if the participants chose to join. All questionnaires were conducted using Google Survey.
4. Interventions The proposed program consisted of eight sessions conducted twice per week, consisting of 5 minutes of introductory material, 12-15 minutes of main content, and 5 minutes of concluding content. The introduction included a brief exercise since exercises can relieve post-traumatic stress symptoms by changing the body's cortisol concentrations (Kim et al., 2013). The main content intended to improve the control processes and each of the four adaptive modes of the Roy Adaptation Model. No session lasted longer than 25 min.

   Participants are given homework and feedback through SNSs. The program's sessions were accessible through blog entries posted on https://www.tistory.com. Every post in the blog required a password. Links and passwords for each session were provided to the participants through SNS. The program was accessible from any electronic device with Internet access, including computers and smartphones, and was strictly accessible through links provided by the researchers.

   The program was partially revised considering the topics' practicality after a feasibility study and consultation with experts.
5. Measurements 1) Trauma experience: Stress Life Events Screening Questionnaire 2) Post-traumatic stress symptoms: Impact of Event Scale-Revised 3) Depression: Center for Epidemiological Studies Depression Scale 4) Functional health: Functional Health Pattern Assessment Screening Tool 5) Adaptation to college life: Students Adjustment to College Questionnaire

ELIGIBILITY:
Inclusion Criteria:

1. female college students between 19 and 29 years
2. who had a traumatic experience
3. who had post-traumatic stress symptom scores of 22-66

Exclusion Criteria:

1. who experienced childhood sexual abuse
2. who had experienced violent conflict or war, including North Korea defectors
3. who had a post-traumatic stress score greater than 66 points

Ages: 19 Years to 29 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Male and female's cognition of trauma is different, and women are vulnerable to post-traumatic stress.
Enrollment: 34 (Actual)
Dates: Start 2020-04-27 (Actual); Primary Completion 2020-11-30 (Actual); Study Completion 2020-12-03 (Actual)

PRIMARY OUTCOMES:
Change of post-traumatic stress symptoms | Baseline, 4 weeks, 8weeks
  Impact of Event Scale-Revised-Korean(IES-R-K). Version for Korean was measured the post traumatic stress symptom of female college students pre-test, post-test 1,2. The total score is 0 ~ 88 points, and the higher the total score, the more severe the post-traumatic stress symptoms.

SECONDARY OUTCOMES:
Change of depression | Baseline, 4 weeks, 8weeks
  Change of depression : Center of Epidemiological Studies Depression Scale (CES-D) Korean version was measured the depression of female college students pre-test, post test 1,2. The total score is 0 ~ 60, and the higher the total score, the more depressed it is.
Fuctional Health | Baseline, 4 weeks, 8weeks
  Functional Health : Functional Health Pattern Assessment Screening Tool (FHPAST) Korean version was measured the functional health of female college students pre-test, post-test 1,2. It consists of a four-point scale (1-4 points), and the higher the score, the better the health function level.
College to adaptation | Baseline, 4 weeks, 8weeks
  College to adaptation : Students Adaptation to College Questionnaire (SACQ). Korean Version was measured the adaptation of college students pre-test, post- test 1,2. It consists of a 9-point scale (1 to 9 points), and the higher the score, the better the adaptation to college life.

CONTACTS AND LOCATIONS:
Overall Officials: Kyunghyun Lee, Ph. D, Principal Investigator — CHA University
Locations (1):
- CHA University, Pocheon-si, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Breslau N, Kessler RC, Chilcoat HD, Schultz LR, Davis GC, Andreski P. Trauma and posttraumatic stress disorder in the community: the 1996 Detroit Area Survey of Trauma. Arch Gen Psychiatry. 1998 Jul;55(7):626-32. doi: 10.1001/archpsyc.55.7.626. PMID 9672053
- [Background] Boyraz G, Horne SG, Owens AC, Armstrong AP. Academic achievement and college persistence of African American students with trauma exposure. J Couns Psychol. 2013 Oct;60(4):582-92. doi: 10.1037/a0033672. Epub 2013 Aug 19. PMID 23957769
- [Background] Kim SH, Schneider SM, Bevans M, Kravitz L, Mermier C, Qualls C, Burge MR. PTSD symptom reduction with mindfulness-based stretching and deep breathing exercise: randomized controlled clinical trial of efficacy. J Clin Endocrinol Metab. 2013 Jul;98(7):2984-92. doi: 10.1210/jc.2012-3742. Epub 2013 May 29. PMID 23720785
- [Background] Knaevelsrud C, Brand J, Lange A, Ruwaard J, Wagner B. Web-based psychotherapy for posttraumatic stress disorder in war-traumatized Arab patients: randomized controlled trial. J Med Internet Res. 2015 Mar 20;17(3):e71. doi: 10.2196/jmir.3582. PMID 25799024
- [Background] Liu H, Petukhova MV, Sampson NA, Aguilar-Gaxiola S, Alonso J, Andrade LH, Bromet EJ, de Girolamo G, Haro JM, Hinkov H, Kawakami N, Koenen KC, Kovess-Masfety V, Lee S, Medina-Mora ME, Navarro-Mateu F, O'Neill S, Piazza M, Posada-Villa J, Scott KM, Shahly V, Stein DJ, Ten Have M, Torres Y, Gureje O, Zaslavsky AM, Kessler RC; World Health Organization World Mental Health Survey Collaborators. Association of DSM-IV Posttraumatic Stress Disorder With Traumatic Experience Type and History in the World Health Organization World Mental Health Surveys. JAMA Psychiatry. 2017 Mar 1;74(3):270-281. doi: 10.1001/jamapsychiatry.2016.3783. PMID 28055082
- [Background] Shipherd JC, Clum G, Suvak M, Resick PA. Treatment-related reductions in PTSD and changes in physical health symptoms in women. J Behav Med. 2014 Jun;37(3):423-33. doi: 10.1007/s10865-013-9500-2. Epub 2013 Mar 8. PMID 23471544
- [Background] Nayback AM. PTSD in the combat veteran: using Roy's Adaptation Model to examine the combat veteran as a human adaptive system. Issues Ment Health Nurs. 2009 May;30(5):304-10. doi: 10.1080/01612840902754404. PMID 19437249
- [Background] Nguyen-Feng VN, Greer CS, Frazier P. Using online interventions to deliver college student mental health resources: Evidence from randomized clinical trials. Psychol Serv. 2017 Nov;14(4):481-489. doi: 10.1037/ser0000154. PMID 29120206
- [Background] Roberts AL, Kubzansky LD, Chibnik LB, Rimm EB, Koenen KC. Association of Posttraumatic Stress and Depressive Symptoms With Mortality in Women. JAMA Netw Open. 2020 Dec 1;3(12):e2027935. doi: 10.1001/jamanetworkopen.2020.27935. PMID 33275156
- [Background] Woods SJ, Isenberg MA. Adaptation as a mediator of intimate abuse and traumatic stress in battered women. Nurs Sci Q. 2001 Jul;14(3):215-21. doi: 10.1177/08943180122108463. PMID 11873342
- [Background] Yehuda R. Post-traumatic stress disorder. N Engl J Med. 2002 Jan 10;346(2):108-14. doi: 10.1056/NEJMra012941. No abstract available. PMID 11784878
- [Background] Seo, Y. S., Jo, H. J., An, H. Y., & Lee, J. S. (2012). Traumatic Events Experenced by South Koreans: Types and Prevalence. Korean journal of counseling and psychotherapy, 24(3), 671-701.
- [Background] Lee, D., Kim, J., & Kim, J. J. (2015). An Exploratory Study on the Possibilities and Limitations of Online Psychotherapy. The Korean Journal of Counseling and Psychotherapy, 27(3), 543-582., Corpus ID: 197667819
- [Background] Lee, K., Jo, H., & Kim, S. (2018). Relationships among Traumatic Experiences, Posttraumatic Stress Symptoms, and Mental Health-related Characteristics in Young Adults. Journal of Korean Academy of Psychiatric and Mental Health Nursing, 27(2), 85. https://doi.org/10.12934/jkpmhn.2018.27.2.85
- [Background] Shin, J., Lee, D.-H., Lee, S.-Y., & Han, Y.-S. (2015). A study on types of traumatic events experienced by undergraduate students. The Journal of Play Therapy, 19(2), 69-95.